CLINICAL TRIAL: NCT06894953
Title: Proof of Concept Study of the Personalised AMPER System (Agent-based Memory Prosthesis to Encourage Reminiscing).
Brief Title: AMPER Proof of Concept Study
Acronym: AMPER
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Strathclyde (Other)
Collaborators: NHS Greater Glasgow and Clyde (Other)
Responsible Party: Principal Investigator, Matt Jamieson, Principal Investigator, University of Strathclyde
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 341144; EP/V05564X/1 (Other Grant/Funding Number: UKRI EPSRC)
Record Dates: First submitted 2025-03-12; First posted 2025-03-25 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Alzheimer's Dementia (AD)
Keywords: Azheimer's disease; Dementia; Reminiscence; Reminiscence technology; Assistive technology; Intelligent Virtual Agent
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Personalised AMPER (Experimental): AMPER app will be provided on a tablet, used with a caregiver in the participant's home for 12 weeks, at least twice a week AND the app will cater topic 'stories' (content) to the persons pre-stated preferences and provide content from the decades that correspond to the person's reminiscence 'bump' (when they were between 10 and 30 years old).
  Interventions: Device: Personalised Agent-based Memory Prosthesis to Encourage Reminiscing (AMPER)
- Non-personalised AMPER (Active Comparator): AMPER app will be provided on a tablet, used with a caregiver in the participant's home for 12 weeks, at least twice a week. AND the app will provide random content not linked to persons preferences or age.
  Interventions: Device: Non-Personalised Agent-based Memory Prosthesis to Encourage Reminiscing (AMPER)

INTERVENTIONS:
Device: Personalised Agent-based Memory Prosthesis to Encourage Reminiscing (AMPER) — AMPER has an embodied agent (CGI character) who will ask questions about various memory cues such as pictures, audio files and videos from a BBC reminiscence archive (https://remarc.bbcrewind.co.uk/) to bring to the surface memories residing in the still viable regions of the brain. Personalised AMPER is personalised to preferences and age of the participant.
  Arms: Personalised AMPER
Device: Non-Personalised Agent-based Memory Prosthesis to Encourage Reminiscing (AMPER) — AMPER has an embodied agent (CGI character) who will ask questions about various memory cues such as pictures, audio files and videos from a BBC reminiscence archive (https://remarc.bbcrewind.co.uk/) to bring to the surface memories residing in the still viable regions of the brain. Non-personliased AMPER is not personalised to preferences or age of the participant.
  Arms: Non-personalised AMPER

SUMMARY:
The AMPER (Agent-based Memory Prosthesis to Encourage Reminiscing) system has been built to help people with Alzheimer's disease by improving their memory recall and quality of life. Alzheimer's often leads to the loss of autobiographical memories, which can affect a person's sense of identity. AMPER seeks to address this by creating a digital memory aid that uses an engaging, animated character on a tablet to help individuals with Alzheimer's reminisce about their past. By presenting personally relevant stories, images, audio, and videos, the character helps trigger memories and encourages interaction with caregivers.

This is proof of concept study using a randomised controlled trial methodology. Twenty participants will be randomised to the control and 20 randomised to the intervention condition. The intervention group will use a personalised version of the AMPER app with tailored content and the control group will use a non-personalised version without specific adaptations. Over 12 weeks, participants will use the app at home with their caregivers. Researchers will measure changes in their memory and cognitive abilities before and after these 12 weeks.

The primary goal is to see if personalised reminiscence improves the perceived quality of the reminiscence experience and autobiographical memory ability compared to the same app with a non-personalised approach. This will be measured using a combination of automatically gathered app use data and weekly caregiver feedback. Secondary goals are to investigate any difference between participants in the intervention and control condition in their technology acceptance, quality of life, self-esteem, everyday functioning and cognitive ability.

Feedback from this research will help refine AMPER and inform future studies, with the ultimate goal of creating a widely accessible tool that supports memory and well-being in Alzheimer's patients. Table 1 provides a summary of the study.

ELIGIBILITY:
Inclusion Criteria:

- Diagnosis of probable Alzheimer's disease of mild to moderate severity according to DSM-IV (Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition) and NINCS-ADRAD (National Institute of Neurological and Communicative Disorders and Stroke-Alzheimer's Disease and Related Disorders Association) criteria.

* Age 50 or older
* Sensory (visual and auditory), language, and physical abilities adequate to perform assessments (corrective aids allowed).
* ACE III score between 20 and 82 (inclusive) (or equivalent score on MMSE (between 14 and 24, based on Law et al., 20123 equivalence data) or MOCHA (between 14 and 24 (based on Pendleberry et al., 2011 equivalence data).
* Having a caregiver or family member who can attend all visits, perform assessments, and supervise administration of study.

Exclusion Criteria:

* Medical records indicate AD patients with the visual variant or having colour vision deficits.
* Medical records indicate a CT or MRI within 24 months prior to screening that indicates a diagnosis other than probable Alzheimer's disease.
* Medical records indicate any significant neurological disease other than probable AD (e.g. Parkinson's disease, Huntington's disease, brain tumor, normal pressure hydrocephalus, progressive supranuclear palsy, seizure disorder, subdural hematoma, multiple sclerosis, history of stroke, or history of head injury requiring hospitalization).
* On review of medical records, no clinically significant abnormal findings on previous physical examination, medical history, or clinical laboratory results that would indicate an alternative diagnosis.
* Current history of major psychiatric disorder (e.g. Major depression) (as indicated on medical records)
* History of substance misuse (as indicated on medical records).

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Quality of autobiographical memory during AMPER use | From enrollment to the end of AMPER use at 12 weeks
  We will analyse the richness of episodic and semantic details in the participant's recollections (which are audio recorded during the trial). This method will ensure a systematic evaluation of memory quality during interactions facilitated by the AMPER app. This rating procedure will use the methodology outlined by Levine and colleagues (2002) and will be scored using the semi-automated methodology outlined by Wardell and colleagues (2021).
Autobiographical Memory ability (objectively rated) | Baseline (week 1) and follow up (week 14)
  Objective rating of Autobiographical Memory ability using the Autobiographical Memory Interview (Kopelman et al., 1989)
Autobiographical Memory ability (subjectively rated) | Baseline (week 1) and follow up (week 14)
  Autobiographical memory ability will be subjectively rated using the Autobiographical Recollection Test (ART), (Berntsen et al., 2019).
Autobiographical Memory ability (subjectively rated on SAM) | Baseline (week 1) and follow up (week 14)
  Autobiographical memory ability will also be subjectively rated using the survey of Autobiographical memory (SAM), (Palombo et al., 2012)

SECONDARY OUTCOMES:
Functional ability in tasks of everyday living | Baseline (week 1) and follow up (week 14)
  Instrumental Activities of Daily Living (IADL), (Lawton & Brody, 1969)
Quality of life for the individual with Alzheimer's disease (subjective) | Baseline (week 1) and follow up (week 14)
  Quality of life Alzheimer's Disease (Logsdon et al., 1999)
Level of Depression experienced by the person with AD (subjective) | Baseline (week 1) and follow up (week 14)
  Geriatric Depression Scale (GDS), (Yesavage et al., 1982),
Cognitive ability of the person with AD | Baseline (week 1) and follow up (week 14)
  Addenbrooke's Cognitive Examination ACE-III (Mioshi et al., 2006)
Verbal learning ability for the person with AD | Baseline (week 1) and follow up (week 14)
  Hopkins Verbal Learning Test (HVLT) (Benedict et al., 1998)
Short term verbal memory for person with AD | Baseline (week 1) and follow up (week 14)
  Digit Span forwards and backwards from the Wechsler Adult Intelligence Scale (4th edition), (Wechsler, 2008)
Executive functioning for person with AD | Baseline (week 1) and follow up (week 14)
  Trail Making Test (Reitan, & Wolfson, 1985)
Modified Hachinski Ischemia Scale score for person with AD | Baseline (week 1) and follow up (week 14)
  Modified Hachinski Ischemia Scale (mHIS) (Hachinski et al., 2012)
Self-esteem for the person with AD | Baseline (week 1) and follow up (week 14)
  The Rosenberg Self Esteem scale (Rosenberg, 1965)
Technology acceptance for person with AD | Baseline (week 1) and follow up (week 14)
  The ALMERE questionnaire (Heerink et al., 2010).

CONTACTS AND LOCATIONS:
Locations (1):
- University of Strathclyde, Glasgow, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided